CLINICAL TRIAL: NCT06366009
Title: Evaluation of the Use of Video EEG Examination Extended With Intra-auricular Electrodes in the Assessment of Patients With Drug-resistant Temporal Lobe Epilepsy
Brief Title: Assessment of Patients With Drug-resistant Temporal Lobe Epilepsy With EEG Extended With Intra-auricular Electrodes
Status: Not yet recruiting | Type: Observational
Sponsor: Przemyslaw Kunert (Industry)
Collaborators: NaoX Technologies (Industry); Warsaw Medical University Clinical Center (Unknown); Departments and Clinics of Emergency Medicine of the Medical University of Gdańsk (Unknown)
Responsible Party: Sponsor-Investigator, Przemyslaw Kunert, Professor Dr. Hab., NaoX Technologies
Organization: NaoX Technologies (Industry)
Other Study IDs: Warsaw Study
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Epilepsy; Focal Epilepsy; Drug Resistant Epilepsy
Keywords: in-ear EEG; EEG; epilepsy; focal epilepsy; drug resistant epilepsy; intra-auricular EEG
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial; Drug Resistant Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: NaoX in-ear EEG system — EEG recordings will be carried out simultaneously using standard EEG equipment (full set of electrodes according to the 10-20 system extended by additional temporal electrodes T9/T10) and the NAOX in-ear EEG system device.
  Other Names: NaoX Buds; standard EEG

SUMMARY:
The study aims to evaluate the effectiveness of long-term video EEG monitoring using 10-20 electrodes extended with intra-auricular electrodes in locating the seizure onset zone and interictal epileptiform discharges (IEDs) in patients with temporal lobe epilepsy (TLE) and nontemporal lobe epilepsy (non-TLE).

DETAILED DESCRIPTION:
This study is a monocentric observational study aiming to evaluate the effectiveness of long-term video EEG monitoring using 10-20 electrodes extended with intra-auricular electrodes in locating the seizure onset zone and interictal epileptiform discharges (IEDs) in patients with temporal lobe epilepsy (TLE) and nontemporal lobe epilepsy (non-TLE).

30 subjects with drug-resistant focal epilepsy undergoing long-term EEG monitoring as part of the pre-surgical assessment will be included.

All patients referred to the UCK WUM Department of Neurosurgery for video EEG monitoring will be subject to prescreening. Those who, according to prior medical documentation, don't meet exclusion criteria and are likely to meet inclusion criteria will be invited to participate in the study and will undergo an initial assessment in form of a structured interview with a clinician, EEG recordings will be carried out simultaneously using standard EEG equipment (full set of electrodes according to the 10-20 system extended by additional temporal electrodes T9/T10) and the NAOX in-ear EEG system device.

EEG monitoring will take place for 5 days of hospitalization according to the standard protocol of the Video-EEG Laboratory of the Department of Neurosurgery, CSK UCK, Medical.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis of drug-resistant epilepsy
* Sufficient level of cooperation to use of the NAOX in-ear EEG system
* Providing informed consent to participate in the study

Exclusion Criteria:

* Presence of skull bone defects, e.g. after prior neurosurgery
* Presence of comorbidities that may significantly affect the resting EEG
* Medical history strongly suggestive of psychogenic nonepileptic attacks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with drug-resistant focal epilepsy undergoing long-term EEG monitoring as part of the pre-surgical assessment.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-04-08 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
determination of the starting point of focal temporal epileptic seizures | Day 5
  correlation of the seizure onset zone encompassing intra-auricular electrodes with the clinically determined location of the focus within the medial temporal lobe

SECONDARY OUTCOMES:
Identification of subgroups of epileptic patterns | Day 5
  Identification of subgroups of epileptic patterns which, depending on the location of the epileptic focus may be more clearly visible at intra-auricular sites than in standard 10-20 system electrode locations, may be visible exclusively at intra-auricular locations, may not be visible at intra-auricular location
Assessment of ease-of-use and comfort of use of the NAOX in-ear EEG system by patients and the EEG technician | Days 1-5
  Questionnaire to EEG technician and patient

CONTACTS AND LOCATIONS:
Locations (1):
- Kliniki Neurochirurgii CSK UCK WUM, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No